CLINICAL TRIAL: NCT00261365
Title: An Exploratory Study to Determine Potential Predictive Markers of Response and/or Toxicity in Patients With Unresectable Stage III or IV Malignant Melanoma Randomized and Treated With Ipilimumab (MDX-010/BMS-734016) at Two Dose Levels
Brief Title: Phase II Study to Determine Predictive Markers of Response to BMS-734016 (MDX-010)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: CA184-004
Record Dates: First submitted 2005-12-01; First posted 2005-12-05 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2008-08

CONDITIONS: Unresectable Stage III or IV Malignant Melanoma
MeSH Terms: interventions — Ipilimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A1 (Active Comparator)
  Interventions: Drug: Ipilimumab
- A2 (Active Comparator)
  Interventions: Drug: Ipilimumab

INTERVENTIONS:
Drug: Ipilimumab — Solution, Intravenous, 3 mg/kg, 3 weeks, 12 - 48 weeks depending on the response.
  Other Names: BMS-734016; (MDX-010)
  Arms: A1
Drug: Ipilimumab — Solution, Intravenous, 10 mg/kg, 3 weeks, 12 - 48 weeks depending on the response.
  Other Names: BMS-734016; (MDX-010)
  Arms: A2

SUMMARY:
The purpose of this study is to identify candidate markers predictive of response and/or serious toxicity to BMS-734016 (MDX-010).

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of unresectable State III or IV malignant melanoma (excluding ocular melanoma); A pre- and post-treatment fresh core or excision tumor biopsy must be provided.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2005-11; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Purpose - to identify candidate markers predictive of response and/or serious toxicity to MDX-101 (BMS-734016) | on a continuous & ongoing basis

SECONDARY OUTCOMES:
Safety & tumor response are important secondary objectives. Safety evaluated | on a continuous & ongoing basis
Tumor response measured | starting @ wk 12 through wk 24. Those continuing on therapy after wk 24 have tumor responses evaluated every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (14):
- United States (3):
  - Comprehensive Cancer Center, Palm Springs, California
  - The Angeles Clinic And Research Institution, Santa Monica, California
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
- Denmark (2):
  - Local Institution, Aarhus C
  - Local Institution, Odense C
- Local Institution, Jerusalem, Israel
- Italy (4):
  - Local Institution, Bari
  - Local Institution, Forlì
  - Local Institution, Ravenna
  - Local Institution, Rimini
- Local Institution, Oslo, Norway
- Local Institution, Lima, Lima Province, Peru
- Sweden (2):
  - Local Institution, Gothenberg
  - Local Institution, Stockholm

REFERENCES:
- [Derived] Schadendorf D, Hodi FS, Robert C, Weber JS, Margolin K, Hamid O, Patt D, Chen TT, Berman DM, Wolchok JD. Pooled Analysis of Long-Term Survival Data From Phase II and Phase III Trials of Ipilimumab in Unresectable or Metastatic Melanoma. J Clin Oncol. 2015 Jun 10;33(17):1889-94. doi: 10.1200/JCO.2014.56.2736. Epub 2015 Feb 9. PMID 25667295
- [Derived] Hamid O, Schmidt H, Nissan A, Ridolfi L, Aamdal S, Hansson J, Guida M, Hyams DM, Gomez H, Bastholt L, Chasalow SD, Berman D. A prospective phase II trial exploring the association between tumor microenvironment biomarkers and clinical activity of ipilimumab in advanced melanoma. J Transl Med. 2011 Nov 28;9:204. doi: 10.1186/1479-5876-9-204. PMID 22123319